CLINICAL TRIAL: NCT05741489
Title: Continuous Glucose Monitoring in Patients With End-Stage Kidney Disease and Burnt-Out Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00004617
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-02

CONDITIONS: End Stage Kidney Disease
Keywords: Burnt-out diabetes; Dialysis; End stage renal disease; Kidney failure
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ESKD with Burnt-out Diabetes (Experimental): Participants with ESKD and burnt-out diabetes wearing a CGM for 10 days.
  Interventions: Device: Continuous glucose monitoring (CGM)
- ESKD without Diabetes (Experimental): Non-diabetic participants with ESKD wearing a CGM for 10 days.
  Interventions: Device: Continuous glucose monitoring (CGM)

INTERVENTIONS:
Device: Continuous glucose monitoring (CGM) — The Dexcom G6 CGM system is a compact, light-weight glucose testing device that measures glucose every 5 minutes. Participants will wear the CGM with the display off for 10 days while continuing their routine dialysis sessions.
  Other Names: Dexcom G6 CGM

SUMMARY:
Twenty participants with end stage kidney disease (ESKD) and burnt-out diabetes, and 20 non-diabetic participants with ESKD will wear a continuous glucose monitoring (CGM) device for 10 days to see if the use of CGM is a better tool to assess glycemic control than glycosylated hemoglobin (HbA1c) in patients with ESKD on dialysis.

DETAILED DESCRIPTION:
More than 37 million adults, or 14.7% of all Americans aged 18 and older, are living with diabetes. Controlling hyperglycemia is foundational to diabetes management and is necessary to reduce the risks of chronic diabetes complications and death. Diabetic nephropathy accounts for great morbidity, as diabetes is the number one cause of chronic kidney disease (CKD) and end stage kidney disease (ESKD) in the United States. It is estimated that diabetes affects up to 40% of patients with ESKD.

Assessment of glucose control in patients with advanced CKD/ESKD is complex due to changes in glucose homeostasis, potential effects on assays of glycemia, and altered pharmacokinetics of diabetes medications. Glycosylated hemoglobin (HbA1c) has been the gold standard to assess glycemic control in patients with diabetes. HbA1c reflects the average glycemic value over approximately 3 months. Although HbA1c is associated with chronic complications of diabetes in patients with normal kidney function, its predictive value is uncertain in patients with ESKD or estimated glomerular filtration rate (eGFR) <30 ml/min. HbA1c reliability in ESKD is reduced because of anemia, shortened erythrocyte lifespan, protein-energy wasting, and malnutrition-inflammation cachexia syndrome, among others. To overcome the limitations of HbA1c, alternative methods to assess long-term glycemic control have been proposed including fructosamine and glycated albumin. Fructosamine measures ketoamines formed by non-enzymatic glycation of serum proteins. It is a useful index for glycemic control over the prior 2 to 4 weeks, and some studies have reported that fructosamine more accurately reflects blood glucose control than HbA1c in anemic patients with ESKD on dialysis. However, there may be falsely low readings in the presence of hypoalbuminemia due to protein-energy wasting and in peritoneal dialysis due to dialysate protein loss. Glycated albumin is a useful marker reflecting glycemic control over the prior 2 to 4 weeks. In patients with ESKD, glycated albumin more rapidly reflects the status of blood glucose control than HbA1c. Like fructosamine, there is potential for falsely low readings in patients with peritoneal dialysis with dialysate protein losses and hypoalbuminemia.

Continuous glucose monitoring (CGM) technology in the outpatient setting has transformed glucose monitoring for diabetes self-management, providing more comprehensive glycemic control data than intermittent point-of-care capillary blood glucose monitoring and HbA1c.

Once progressed to ESKD, up to one fourth of patients experience resolution of their hyperglycemia, as defined by an HbA1c level of less than 6.5%, and consequently are no longer on antidiabetic agents and insulin. This phenomenon is known as "burnt-out diabetes" which is likely due to various underlying factors, including but not limited to, malnutrition, reduced clearance and degradation of insulin, decreased kidney gluconeogenesis, and accumulation of uremic toxins. These patients are likely at a greater risk of morbidity and mortality and an increased risk of hypoglycemic episodes. There is a need for further research in patients with ESKD to establish what is the most appropriate tool to assess glycemic control in those with 'burnt-out diabetes'.

This study will use CGM to measure patients' glucose with real-time levels as opposed to relying on surrogate markers like HbA1c. These results can give insight into the reality of glycemic control in these patients and can impact the best monitoring and treatment for patients with burnt-out diabetes. It is not known if patients with burnt-out diabetes have complete normoglycemia or if they may have episodes of (untreated) hyperglycemia, which may be associated with poor outcomes. The researchers of this study will compare glycemic control by CGM in patients with burnt-out diabetes and non-diabetic patients with ESKD.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis treatment for more than 3 months
* HbA1c less than 6.5% at the first clinic visit
* Willing to wear a CGM for 10 days

Exclusion Criteria:

* Have used insulin or any diabetes treatment during the last 3 months
* Be pregnant or plan to become pregnant during the study
* Known allergy to medical-grade adhesives
* Taking acetaminophen (more than 1 gram every six hours) or hydroxyurea (may interfere with sensor membrane)
* Current or anticipated use of stress steroid doses (prednisone </= 5 mg or its equivalent is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory Dialysis at Northside, Atlanta, Georgia
  - Emory Dialysis at Greenbriar, Atlanta, Georgia
  - Emory Dialysis at Candler, Decatur, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kaminski CY, Galindo RJ, Navarrete JE, Zabala Z, Moazzami B, Gerges A, McCoy RG, Fayfman M, Vellanki P, Idrees T, Peng L, Umpierrez GE. Assessment of Glycemic Control by Continuous Glucose Monitoring, Hemoglobin A1c, Fructosamine, and Glycated Albumin in Patients With End-Stage Kidney Disease and Burnt-Out Diabetes. Diabetes Care. 2024 Feb 1;47(2):267-271. doi: 10.2337/dc23-1276. PMID 38085705

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Emory Dialysis centers in Atlanta, Georgia, USA. Participant enrollment began August 10, 2022 and all follow-up assessments were completed by March 9, 2023.
Groups:
- End-Stage Kidney Disease (ESKD) With Burnt-out Diabetes: Participants with end stage kidney disease (ESKD) and burnt-out diabetes wearing a continuous glucose monitoring (CGM) for 10 days. The Dexcom G6 CGM system is a compact, light-weight glucose testing device that measures glucose every 5 minutes. Participants wore the CGM with the display off for 10 days while continuing their routine dialysis sessions.
- ESKD Without Diabetes: Non-diabetic participants with ESKD wearing a CGM for 10 days. The Dexcom G6 CGM system is a compact, light-weight glucose testing device that measures glucose every 5 minutes. Participants wore the CGM with the display off for 10 days while continuing their routine dialysis sessions.
Period: Overall Study
Arm/Group | End-Stage Kidney Disease (ESKD) With Burnt-out Diabetes | ESKD Without Diabetes
Started | 20 | 20
Completed | 20 | 18
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- ESKD With Burnt-out Diabetes: Participants with ESKD and burnt-out diabetes wearing a CGM for 10 days. The Dexcom G6 CGM system is a compact, light-weight glucose testing device that measures glucose every 5 minutes. Participants wore the CGM with the display off for 10 days while continuing their routine dialysis sessions.
- Total: Total of all reporting groups
Arm/Group | ESKD With Burnt-out Diabetes | ESKD Without Diabetes | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.3) | 60.1 (9.5) | 61.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 10 | 12 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 20 | 40
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40
Coronary artery disease [Count of Participants; unit: Participants] | 7 | 3 | 10
Heart failure [Count of Participants; unit: Participants] | 14 | 15 | 29
Hypertension [Count of Participants; unit: Participants] | 20 | 18 | 38
Hemoglobin A1c (HbA1c) [Count of Participants; unit: Participants]
  < 5.7% | 10 | 13 | 23
  5.7 to < 6.5% | 10 | 7 | 17
Glycated albumin level [Count of Participants; unit: Participants]
  less than 13.6% | 2 | 7 | 9
  13.6% to < 16% | 4 | 5 | 9
  greater than or equal to 16% | 12 | 6 | 18
  not assessed | 2 | 2 | 4
Fructosamine level (mmol/L) [Count of Participants; unit: Participants]
  less than 285 | 3 | 5 | 8
  greater than or equal to 285 | 15 | 13 | 28
  not assessed | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent of Time in Range (TIR) Between 70-180 mg/dL
Description: Glycemic control is measured as the percentage of time that blood glucose levels are in the range of 70 and 180 mg/dL, as measured by CGM.
Time Frame: Up to 10 days
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | ESKD With Burnt-out Diabetes | ESKD Without Diabetes
Number analyzed (Participants) | 20 | 18
percentage of time | 80.4 (14.0) | 94.0 (6.4)

2. Primary Outcome: Percent of Time Above Range (Blood Glucose >180 mg/dL)
Description: Glycemic control is assessed a the percentage of time in hyperglycemia, defined as the time above range (TAR) with blood glucose measurements >180 mg/dL, as measured by CGM.
Time Frame: Up to 10 days
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | ESKD With Burnt-out Diabetes | ESKD Without Diabetes
Number analyzed (Participants) | 20 | 18
percentage of time | 17.2 (14.1) | 4.6 (5.3)

3. Primary Outcome: Percent of Time Above Range (Blood Glucose >250 mg/dL)
Description: Glycemic control is assessed a the percentage of time in hyperglycemia, defined as the time above range (TAR) with blood glucose measurements >250 mg/dL, as measured by CGM.
Time Frame: Up to 10 days
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | ESKD With Burnt-out Diabetes | ESKD Without Diabetes
Number analyzed (Participants) | 20 | 18
percentage of time | 2.0 (3.0) | 0.1 (0.4)

4. Primary Outcome: Duration of Hyperglycemia (Blood Glucose >180 mg/dL)
Description: Glycemic control is assessed as the duration of hyperglycemia with blood glucose measurements >180 mg/dL, as measured by CGM for hyperglycemia time periods of greater than 15 minutes.
Time Frame: Up to 10 days
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | ESKD With Burnt-out Diabetes | ESKD Without Diabetes
Number analyzed (Participants) | 20 | 18
hours per day | 4.1 (3.4) | 1.1 (1.3)

5. Primary Outcome: Duration of Hyperglycemia (Blood Glucose >250 mg/dL)
Description: Glycemic control is assessed as the duration of hyperglycemia with blood glucose measurements >250 mg/dL, as measured by CGM for hyperglycemia time periods of greater than 15 minutes.
Time Frame: Up to 10 days
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | ESKD With Burnt-out Diabetes | ESKD Without Diabetes
Number analyzed (Participants) | 20 | 18
hours per day | 0.5 (0.7) | 0.1 (0.1)

6. Primary Outcome: Number of Participants With Hyperglycemic Episodes With Blood Glucose >250 mg/dL
Description: The number of participants experiencing hyperglycemia with blood glucose levels > 250 mg/dL as measured by CGM.
Time Frame: Up to Day 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESKD With Burnt-out Diabetes | ESKD Without Diabetes
Number analyzed (Participants) | 20 | 18
Participants | 11 | 3

7. Primary Outcome: Percent of Time Below Range (Blood Glucose <70 mg/dL)
Description: Glycemic control is assessed a the percentage of time in hypoglycemia, defined as the time below range (TBR) with blood glucose measurements < 70 mg/dL, as measured by CGM.
Time Frame: Up to 10 days
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | ESKD With Burnt-out Diabetes | ESKD Without Diabetes
Number analyzed (Participants) | 20 | 18
percentage of time | 2.5 (5.8) | 1.5 (5.0)

8. Primary Outcome: Percent of Time Below Range (Blood Glucose <54 mg/dL)
Description: Glycemic control is assessed a the percentage of time in severe hypoglycemia, defined as the time below range (TBR) with blood glucose measurements < 54 mg/dL, as measured by CGM.
Time Frame: Up to 10 days
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | ESKD With Burnt-out Diabetes | ESKD Without Diabetes
Number analyzed (Participants) | 20 | 18
percentage of time | 1.3 (3.5) | 0.4 (1.7)

9. Primary Outcome: Hypoglycemia Event Rate
Description: Hypoglycemia is defined as blood glucose < 70 mg/dL and is assessed by Dexcom G6 CGM. The hypoglycemic event rate is defined as the number of hypoglycemic events per patient per day.
Time Frame: Up to Day 10
Measure: Mean (Standard Deviation); unit: events per patient per day
Arm/Group | ESKD With Burnt-out Diabetes | ESKD Without Diabetes
Number analyzed (Participants) | 20 | 18
events per patient per day | 3.60 (7.37) | 3.44 (10.43)

10. Primary Outcome: Number of Participants With Hypoglycemic Episodes
Description: The number of participants experiencing hypoglycemia with blood glucose levels < 70 mg/dL as measured by CGM.
Time Frame: Up to Day 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESKD With Burnt-out Diabetes | ESKD Without Diabetes
Number analyzed (Participants) | 20 | 18
Participants | 10 | 11

11. Primary Outcome: Nocturnal Hypoglycemia Event Rate
Description: Hypoglycemia is defined as blood glucose < 70 mg/dL and is assessed by Dexcom G6 CGM. A nocturnal hypoglycemia episode is defined as an episode occurring during the time interval of 10:00 Post Meridiem (PM) to 6:00 Ante Meridiem (AM). The hypoglycemic event rate is defined as the number of hypoglycemic events per patient per day.
Time Frame: Up to Day 10
Measure: Mean (Standard Deviation); unit: events per patient per day
Arm/Group | ESKD With Burnt-out Diabetes | ESKD Without Diabetes
Number analyzed (Participants) | 20 | 18
events per patient per day | 1.30 (3.05) | 0.94 (2.86)

12. Primary Outcome: Number of Participants With Nocturnal Hypoglycemic Episodes
Description: The number of participants experiencing nocturnal hypoglycemia with blood glucose levels < 70 mg/dL as measured by CGM. A nocturnal hypoglycemia episode is defined as an episode occurring during the time interval of 10:00 Post Meridiem (PM) to 6:00 Ante Meridiem (AM).
Time Frame: Up to Day 10
Measure: Count of Participants; unit: Participants
Arm/Group | ESKD With Burnt-out Diabetes | ESKD Without Diabetes
Number analyzed (Participants) | 20 | 18
Participants | 7 | 4

13. Secondary Outcome: Mean Daily Blood Glucose Concentration
Description: Glycemic control is assessed as mean daily glucose concentration, measured by Dexcom G6 CGM.
Time Frame: Up to Day 10
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ESKD With Burnt-out Diabetes | ESKD Without Diabetes
Number analyzed (Participants) | 20 | 18
mg/dL | 141.7 (22.2) | 125.7 (13.7)

14. Secondary Outcome: Glycemic Variability Calculated by Mean Amplitude of Glycemic Excursions (MAGE)
Description: Mean amplitude of glycemic excursions (MAGE) is the parameter for assessing glycemic variability and is calculated based on the arithmetic mean of differences between consecutive peaks and nadirs of differences greater than one standard deviation (SD) of mean glucose values. It is designated to assess major glucose swings and exclude minor ones.
Time Frame: Up to 10 Days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ESKD With Burnt-out Diabetes | ESKD Without Diabetes
Number analyzed (Participants) | 20 | 18
mg/dL | 54.9 (18.2) | 42.4 (9.4)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time individuals gave consent to participate in the study and continued up to Day 10.
Arm/Group | ESKD With Burnt-out Diabetes | ESKD Without Diabetes
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/89/NCT05741489/Prot_SAP_000.pdf